CLINICAL TRIAL: NCT06968429
Title: Efficacy and Safety of Oral NBP Soft Capsules for the Prevention of Episode Migraine Attacks in Adult Migraine Patients: a Multi-center, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Oral NBP Soft Capsules for the Prevention of Episode Migraine Attacks in Adult Migraine Patients
Acronym: ENERGY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University First Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The People's Hospital of Hebei Province (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Dong, MD, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2024-399-02; 2023YFC2508703 (Other Grant/Funding Number: The National Key Research and Development Program of China)
Record Dates: First submitted 2025-04-21; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP (Experimental)
  Interventions: Drug: NBP Softgel Capsules
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBP Softgel Capsules — take orally on an empty stomach；2 capsules 3/day
  Arms: NBP
Drug: Placebo — take orally on an empty stomach；2 capsules 3/day
  Arms: placebo

SUMMARY:
This is a multicentre, randomised, double-blind, placebo-controlled study to evaluate the efficacy, safety and tolerability of oral butylphthalide soft capsules for the prophylactic treatment of migraine in adults.

ELIGIBILITY:
Only patients who meet all of the following criteria will be enrolled in this study:

A history of migraine (with or without aura) for at least 1 year according to the diagnostic criteria of the ICHD-3 and the following criteria:

* Age of onset of migraine before 50 years of age
* If untreated, the average migraine attack lasts 4-72 hours
* 4-14 days of migraine attacks per month in the 3 months prior to the screening visit, as reported by the subject
* at least 4 or more migraine days during the 28-day observation period, according to headache diaries
* No more than 14 headache days within the 28-day observation period according to headache diary
* Ability to differentiate between migraine attacks and tension/cluster headaches

Reproductive status:

* Women of childbearing potential (WOCBP) and non-sterilised men must use an acceptable method of contraception throughout the study period to minimise the risk of pregnancy
* For men undergoing vasectomy, they are considered surgically sterilised if the procedure was performed prior to 6 months (24 weeks) of their participation in the study

Patient compliance:

* Headache diary reports must be completed for at least 24 days during the 28-day observation period
* Subjects must be able to read, understand and complete the study questionnaire and headache diary, at the investigator's discretion

No clinically significant abnormalities are present:

* No clinically significant abnormality found by medical or laboratory evaluation
* Subjects presenting with clinical abnormalities or laboratory parameters outside of reference ranges may be included in the study if the investigator believes that these findings are not clinically significant, do not introduce additional risk factors, and do not interfere with the study procedures

Exclusion Criteria:

Patients will be excluded from this study if they meet any of the following criteria:

Target Disease Exclusion:

* Migraine with brainstem aura or hemiplegic migraine
* Headache (migraine or non-migraine) ≥ 15 days per month in any month during the 3 months prior to the screening visit
* Patients with migraine with medication overuse headache

Medical history and co-morbidities:

* History of HIV infection
* Migraine or head or neck regional interventions/devices (e.g., nerve blocks or transcranial magnetic stimulation) within 2 months prior to enrolment
* Uncontrolled, unstable or recently diagnosed cardiovascular disease (ischaemic heart disease, coronary vasospasm and cerebral ischaemia). Myocardial infarction, acute coronary syndrome, undergoing percutaneous coronary intervention, cardiac surgery, experiencing a stroke or transient ischaemic attack within 6 months (24 weeks) prior to the screening visit.
* Uncontrolled hypertension or uncontrolled diabetes mellitus. Subjects with a history of hypertension, hypercholesterolaemia and/or diabetes mellitus but whose current status is stable and controlled and who have been receiving a stable dose of medication for at least 3 months (12 weeks) prior to the Screening Visit may be enrolled in the study.
* History of gastric or small bowel surgery (including gastric bypass, gastric banding, sleeve gastrectomy, intragastric ballooning, etc.) or a condition that causes malabsorption (e.g., chronic pancreatitis, ulcerative colitis, etc.)
* History of Gilbert's syndrome or current diagnosis of Gilbert's syndrome or any other active liver or biliary tract disease.
* Diagnosis of haematological or solid malignancy within 5 years prior to screening. For subjects with a history of localised basal cell carcinoma or squamous cell skin cancer, they will be eligible to participate in this study if they are confirmed to be cancer free prior to the screening visit.
* Any previous or current unstable medical condition (e.g., congenital heart disease or history of cardiac arrhythmia, known or suspected infection, cancer) that, in the opinion of the investigator, would place the subject at increased risk of a significant adverse event during the course of the trial or interfere with the safety/efficacy assessment.
* Active chronic pain syndromes (e.g. fibromyalgia, chronic pelvic pain, complex localised pain syndrome).
* Have other pain syndromes (including trigeminal neuralgia), psychiatric disorders, dementia, or major neurological disorders (other than migraine) that, in the opinion of the investigator, may interfere with study evaluation
* Current or previous diagnosis of schizophrenia, bipolar disorder or borderline personality disorder
* Has had a depressive episode within the past 12 months or requires more than 1 standard treatment medication daily to treat their depressive disorder or anxiety disorder. For medications used to treat a depressive disorder or anxiety disorder, the medication must have been maintained at a stable dose for at least 3 months prior to the Screening Visit.
* History, treatment history, or evidence of alcohol or drug abuse in the 12 months (48 weeks) prior to the Screening Visit, or a history of substance abuse consistent with any of the DSM-5 Significant Substances in the 12 months (48 weeks) prior to the Screening Visit through the end of the double-blind treatment period.
* Subjects should be excluded if they have a positive screening result for addictive drugs that, in the opinion of the Investigator, is medically significant and would compromise the safety of the subject or the interpretation of the study results. In addition:
* Cocaine, amphetamines, phencyclidine (PCP), and tetrahydrocannabinol (THC) at detectable levels on the Drug Screen need to be excluded.
* Subjects who have a positive drug screen for amphetamines and are using a prescription amphetamine drug for one of the approved indications (e.g., Attention Deficit Hyperactivity Disorder [ADHD]) may be enrolled in the study at the discretion of the Investigator. The Investigator's decision must be documented in detail in the subject's source medical record. Stimulant dosage must remain stable from the first 3 months (12 weeks) of the observation period to the end of the double-blind treatment period.
* BMI ≥ 33.0 kg/m2

ECG and laboratory findings:

* Corrected QT interval > 470 ms at screening (QTc corrected using the Fridericia method)
* left bundle branch block
* Right bundle branch block with QRS duration ≥150 ms
* Intracardiac conduction defect with QRS duration ≥150 ms
* Serum bilirubin (total bilirubin, direct bilirubin, or indirect bilirubin) > 2 x ULN.
* AST or ALT > 3 × ULN.
* Neutrophil count ≤ 1000/μL (or equivalent)

Allergies and other factors:

* History of celery allergy
* Tendency to bleed

Reproductive status:

* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception or abstinence to avoid pregnancy throughout the study period and for 60 days after the last dose of study drug.
* Females who are pregnant or breastfeeding.
* Females with a positive pregnancy test result at screening or prior to study drug administration.

Men of childbearing potential who have an active sex life with a woman of childbearing potential but are unwilling or unable to use one or more acceptable methods of contraception or abstinence to avoid pregnancy with their partner throughout the study period and for 90 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The change of the average monthly migraine days after treatment | Baseline and weeks 12
  The changes of migraine days each month compared with the observation period throughout the double-blind treatment period (weeks 1 to 12).

SECONDARY OUTCOMES:
The change in the frequency of using acute painkillers | Baseline and weeks 12
  The change in the average monthly days of using any acute headache medication 12 weeks after the first administration of butylphthalide soft capsules relative to the observation period

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared in the website of SESH: https://www.seshglobal.org/, within 6 months after the end of research.
URL: https://www.seshglobal.org/